CLINICAL TRIAL: NCT06272786
Title: The Effect of Suprascapular Nerve Block in Patients Rehabilitated After Arthroscopic Rotator Cuff Repair: Randomized Controlled Study
Brief Title: Suprascapular Nerve Block in Patients Rehabilitated After Arthroscopic Rotator Cuff Repair
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Basak Cigdem Karacay, Principal Investigator, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-18/128
Record Dates: First submitted 2024-02-13; First posted 2024-02-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Rotator Cuff Tears; Pain; Nerve Block
Keywords: Rotator Cuff Tears; pain; nerve block; rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Pain

STUDY DESIGN:
Intervention Model Description: Randomised controlled
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcome assessor will be different persons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In addition to the conventional physiotherapy program, patients in the intervention group will receive a suprascapular nerve block with musculoskeletal USG guidance available in our clinic at the beginning of rehabilitation. Bupivacaine hydrochloride will be used in this injection. 5 ml of bupivacaine hydrochloride 5% and 5 ml of saline will be drawn into a 10 ml syringe and ejection will be performed from the superior of the suprascapular noch under USG guidance.
  Interventions: Procedure: conventional physiotherapy program.; Procedure: Suprascapular nerve block
- Control Group (Active Comparator): Patients in the control group will only receive a conventional physiotherapy program.
  Interventions: Procedure: conventional physiotherapy program.

INTERVENTIONS:
Procedure: conventional physiotherapy program. — It will be applied to a rehabilitation program including joint range of motion exercises and physical therapy modalities by a physiotherapist at the Physical Therapy Hospital.
Procedure: Suprascapular nerve block — Bupivacaine hydrochloride will be used in this injection. 5 ml of bupivacaine hydrochloride 5% and 5 ml of saline will be drawn into a 10 ml syringe and ejection will be performed from the superior of the suprascapular noch under USG guidance.
  Arms: Experimental Group

SUMMARY:
Suprascapular nerve block is an injection method that has been shown to be effective in shoulder rehabilitation in diseases such as adhesive capsulitis and stroke .. Applying the block under USG guidance instead of blinding increases the effectiveness and reduces complications.

DETAILED DESCRIPTION:
Suprascapular nerve block is an injection method that has been shown to be effective in shoulder rehabilitation in diseases such as adhesive capsulitis and stroke .Applying the block under USG guidance instead of blinding increases the effectiveness and reduces complications There are many studies in the literature on suprascapular, axillary, and interscalene nerve blocks in early pain management after shoulder arthroplasty. All of these focus on pain in the perioperative or early postoperative period. There is a study on USG-guided suprascapular nerve block. In this study, unlike the studies in the literature, it was aimed to show the effectiveness of USG-guided suprascapular nerve block in the subacute rehabilitation process of patients.

ELIGIBILITY:
Inclusion Criteria:

-Having undergone arthroscopic rotator cuff repair surgery within the last week

Exclusion Criteria:

* History of previous surgery on the same shoulder
* History of systemic inflammatory rheumatological disease
* Neurological diseases with muscle weakness in the upper extremity (MS, ALS, Muscular -Dystrophy)
* History of malignancy, pregnancy, breastfeeding
* Use of steroids or immunosuppressive drugs
* History of allergic reactions to local analgesics
* Fibromyalgia syndrome
* Chronic painful conditions that require opioid use
* Presence of known psychiatric disease
* Cognitive impairment (Mini Mental Test Score <23)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-28 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline
  In the study, pain intensity was evaluated with the Visual Analogue Scale (VAS). Numbers from 0 to 10 on VAS; Patients will be asked to score their pain levels at rest, activity and at night, with 0 being defined as "no pain" and 10 being "unbearable pain". Increased scores indicate higher pain intensity.
Visual Analog Scale (VAS) | 6th week
  In the study, pain intensity was evaluated with the Visual Analogue Scale (VAS). Numbers from 0 to 10 on VAS; Patients will be asked to score their pain levels at rest, activity and at night, with 0 being defined as "no pain" and 10 being "unbearable pain". Increased scores indicate higher pain intensity.
Visual Analog Scale (VAS) | 10th week
  In the study, pain intensity was evaluated with the Visual Analogue Scale (VAS). Numbers from 0 to 10 on VAS; Patients will be asked to score their pain levels at rest, activity and at night, with 0 being defined as "no pain" and 10 being "unbearable pain". Increased scores indicate higher pain intensity.
Shoulder joint range of motion (ROM) | Baseline
  Joint range of motion will be measured and recorded passively in all directions using a goniometer according to the neutral zero method.
Shoulder joint range of motion (ROM) | 6th week
  Joint range of motion will be measured and recorded passively in all directions using a goniometer according to the neutral zero method.
Shoulder joint range of motion (ROM) | 10 th week
  Joint range of motion will be measured and recorded passively in all directions using a goniometer according to the neutral zero method.

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index (SPADİ) | Baseline
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. The score of the total and all sub-parameters is evaluated on a scale of 0-100. A high score indicates increased pain and impaired shoulder function.
Shoulder Pain and Disability Index (SPADİ) | 6th week
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. The score of the total and all sub-parameters is evaluated on a scale of 0-100. A high score indicates increased pain and impaired shoulder function.
Shoulder Pain and Disability Index (SPADİ) | 10th week
  SPADI is a scale consisting of a total of 13 questions with 2 subscales: pain and disability. The score of the total and all sub-parameters is evaluated on a scale of 0-100. A high score indicates increased pain and impaired shoulder function.
Modified Constant-Murley Scoring | 6th week
  Modified Constant-Murley Scoring includes a total of four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a scale of 0-100 points by summing all subparametricS. A low score reflects increased pain and impaired shoulder functions, both in terms of subparametrics and the total score.
Modified Constant-Murley Scoring | 10th week
  Modified Constant-Murley Scoring includes a total of four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a scale of 0-100 points by summing all subparametricS. A low score reflects increased pain and impaired shoulder functions, both in terms of subparametrics and the total score.
Modified Constant-Murley Scoring | Baseline
  Modified Constant-Murley Scoring includes a total of four parameters: pain, activities of daily living (ADL), active ROM and strength. The total score is evaluated on a scale of 0-100 points by summing all subparametricS. A low score reflects increased pain and impaired shoulder functions, both in terms of subparametrics and the total score.

CONTACTS AND LOCATIONS:
Overall Officials: Basak Cigdem Karacay, Asst Prof, Principal Investigator — Kirsehir Ahi Evran University
Locations (1):
- Ahi Evran University, Kirşehir, City Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No